CLINICAL TRIAL: NCT02081586
Title: mHealth Skill Enhancement Plus Phone CBT for Type 2 Diabetes Distress Medication Nonadherence: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Judith A. Callan PhD. RN, Research Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO13040441; KL2TR000146 (NIH)
Record Dates: First submitted 2014-03-03; First posted 2014-03-07 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: CBT; Type 2 Diabetes; Diabetes Distress; Adherence; Smartphone App; Self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 6 Weeks Phone CBT plus smartphone app (Experimental): Following baseline, six 30-minute sessions of phone CBT to address any beliefs, assumptions, attitudes, or perceptions that are not constructive to diabetes self-management. CBT phone app will assist patients to practice skills related to improving self-management via more constructive ways of thinking.
  Interventions: Behavioral: CBT; Device: Smartphone app; Other: Standard Diabetes Care at PCP
- 8 Weeks Phone CBT plus smartphone app (Experimental): Following baseline, patients will receive 8 weeks of phone CBT to address non-constructive beliefs, assumptions, attitudes or perceptions related to diabetes self-management. They will have a smartphone apps to practice CBT skills between sessions.
  Interventions: Behavioral: CBT; Device: Smartphone app; Other: Standard Diabetes Care at PCP
- 12 weeks phone CBT plus smartphone app (Experimental): Following baseline, patients will receive 12 weeks of phone CBT to address non-constructive beliefs, assumptions, attitudes or perceptions related to diabetes self-management. They will have a smartphone apps to practice CBT skills between sessions.
  Interventions: Behavioral: CBT; Device: Smartphone app; Other: Standard Diabetes Care at PCP
- Standard Diabetes Care at PCP (Active Comparator): Patients will remain in usual care and not receive study intervention. This will include usual diabetes care at PCP.
  Interventions: Other: Standard Diabetes Care at PCP

INTERVENTIONS:
Behavioral: CBT — Therapists will work with patients to identify non-constructive thinking patterns that are serving as barriers to adequate self-management of Type 2 Diabetes.
  Other Names: Cognitive Behavioral Therapy
  Arms: 12 weeks phone CBT plus smartphone app; 6 Weeks Phone CBT plus smartphone app; 8 Weeks Phone CBT plus smartphone app
Device: Smartphone app — Smartphone app developed to assist patients practice CBT skills throughout the week
  Other Names: CBT Mobile Work
  Arms: 12 weeks phone CBT plus smartphone app; 6 Weeks Phone CBT plus smartphone app; 8 Weeks Phone CBT plus smartphone app
Other: Standard Diabetes Care at PCP — Patients receive ADA standard of Care with physician at PCP office

SUMMARY:
This is a pilot study examining the clinical effects of a brief Cognitive Therapy phone approach augmented with a CBT smartphone app geared towards patients with type 2 diabetes patients in poor control.

DETAILED DESCRIPTION:
A significant problem in primary care healthcare delivery is the lack of interventions to improve medication and overall regimen adherence in persons with Type 2 diabetes (T2DM). Diabetes distress, a negative response to the diagnosis of T2DM, danger of complications, and self-management burdens is present in up to 70% of persons with T2DM. Distress is a significant factor in medication nonadherence and poor glycemic control. Treatment adherence is vital to maintain glucose control and reduce complications.

The literature has identified dysfunctional thinking patterns such as beliefs (e.g., I can't handle taking these medications), assumptions (e.g., I know I will have side effects to these medications) and interpretations (e.g., I'm too overwhelmed to do all of this stuff) as critical variables that impact both distress and T2DM treatment adherence. Current treatment strategies within primary care do not address the dysfunctional thinking patterns that affect the patient's distress level, T2DM medication adherence, and complex daily self-care activities.

Cognitive behavior therapy (CBT), a well-established evidenced-based treatment, helps patients to identify, and restructure dysfunctional thinking patterns. The investigators propose to test a brief phone CBT approach that is supported by a comprehensive mobile phone CBT skills practice application (app) within primary care. The promising results of the investigators preliminary studies using a mobile phone app to stimulate real-time CBT skills practice prompt us to propose a pilot of its use with patients with T2DM with the following aims:

Primary aim: examine feasibility and acceptability of the assessment protocol, and the recruitment, and retention of study participants.

Secondary aim: 1) collect preliminary data on the effect of the intervention on clinical outcomes, e.g., self-reported adherence to medication and self-management adherence, e.g., diet, exercise; levels of diabetes distress, diabetes medication beliefs, and distal T2DM outcomes (HbA1c level and body mass index).

ELIGIBILITY:
Inclusion Criteria:

1. have a diagnosis of T2DM;
2. have a score of >3 on the Diabetes Distress Scale;
3. be taking at least one oral antihyperglycemic agent (the patient may also be using injectable antihyperglycemic medications, including insulin);
4. have an HbA1c level of greater than 8 at baseline;
5. be receiving treatment for T2DM in the primary care setting;
6. be aged 30 - 65 years and
7. be able to read at the 8th-grade level and to provide informed consent. -

Exclusion Criteria:

1. diagnosis of bipolar disorder or schizophrenia; primary diagnosis of obsessive-compulsive disorder, posttraumatic stress disorder, substance abuse, or dependence in the last 6 months; or any psychotic disorder;
2. diabetes treated without oral medications;
3. inability to read or comprehend English at the 8th-grade level;
4. refusal to provide informed consent;
5. dementia or disorders with substantial cognitive impairment; and
6. serious suicidal risk -

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Callan, PhD, Principal Investigator — University of Pittsburgh School of Nursing
Locations (1):
- University of Pittsburgh School of Nursing, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Callan JA, Sereika SM, Cui R, Tamres LK, Tarneja M, Greene B, Van Slyke A, Wu M, Lukac GR, Dunbar-Jacob J. Cognitive Behavioral Therapy (CBT) Telehealth Augmented With a CBT Smartphone Application to Address Type 2 Diabetes Self-Management: A Randomized Pilot Trial. Sci Diabetes Self Manag Care. 2022 Dec;48(6):492-504. doi: 10.1177/26350106221133027. Epub 2022 Nov 9. PMID 36350066

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment as Usual: Patients will remain in usual care and not receive study intervention.
  Standard Diabetes Care at PCP: Patients receive ADA standard of Care with physician at PCP office
Period: Overall Study
Arm/Group | 6 Weeks Phone CBT Plus Smartphone App | 8 Weeks Phone CBT Plus Smartphone App | 12 Weeks Phone CBT Plus Smartphone App | Treatment as Usual
Started | 3 | 3 | 4 | 3
Completed | 3 | 2 | 3 | 2
Not Completed | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Head injury not related to study | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 Weeks Phone CBT Plus Smartphone App | 8 Weeks Phone CBT Plus Smartphone App | 12 Weeks Phone CBT Plus Smartphone App | Treatment as Usual | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (1.0) | 50.67 (12.34) | 59.50 (3.42) | 60.67 (.58) | 57.38 (6.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 3 | 9
  Male | 2 | 1 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 1 | 1 | 7
  White | 0 | 1 | 3 | 2 | 6
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Level Change Scores From Baseline to 16 Weeks
Description: Change from baseline HbA1c level to post intervention
Time Frame: baseline to 16 weeks
Population: per protocol
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | 6 Weeks Phone CBT Plus Smartphone App | 8 Weeks Phone CBT Plus Smartphone App | 12 Weeks Phone CBT Plus Smartphone App | Treatment as Usual
Number analyzed (Participants) | 3 | 2 | 3 | 2
percent | -0.60 (.26) | -2.30 (.00) | -2.33 (.50) | -2.15 (1.63)

2. Primary Outcome: Computer System Usability Questionnaire (CSUQ)
Description: The CSUQ measures feasibility and acceptability of the phone application. Adapted from Lewis JR.: IBM Computer Usability Satisfaction Questionnaires: Psychometric Evaluation and Instructions for Use. International Journal of Human-Computer Interaction 1995; 7 (1):67-78.
  Scale is scored as a mean value, range is from 1 to 7. In this adaptation lower scores are better usability.
Time Frame: 16 weeks
Population: As per protocol, usability was analyzed for participants administered phone CBT, regardless of duration. Six subjects completed the CSUQ. Of ten initially assigned treatment, one was withdrawn prior to treatment, one missed the CSUQ, and two dropped out. Treatment as usual Arm did not use the phone.
Measure: Mean (Standard Deviation); unit: units on a scale (1-7)
Groups:
- Participants Administered Phone CBT: This includes the 3 treatment arms who received Phone CBT, whether CBT treatment was 6, 8, or 12 weeks long.
Arm/Group | 6 Weeks Phone CBT Plus Smartphone App | 8 Weeks Phone CBT Plus Smartphone App | 12 Weeks Phone CBT Plus Smartphone App | Treatment as Usual | Participants Administered Phone CBT
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6
units on a scale (1-7) |  |  |  |  | 3.0 (2.1)

3. Secondary Outcome: MEMS (Medication Electronic Monitoring System) Cap Electronic Pill Bottle Adherence
Description: Electronically measured medication adherence, percent adherence over entire study phase. Change score was not evaluated, this measure is to determine feasability of use over time. Percent adherence is measured by the number of correct doses per day divided by the number of prescribed doses per day X 100. Percent adherence was calculated as the percentage of the prescribed doses of the medication actually taken by the patient over 16 weeks
Time Frame: 16 weeks
Measure: Mean (Full Range); unit: percent adherent
Arm/Group | 6 Weeks Phone CBT Plus Smartphone App | 8 Weeks Phone CBT Plus Smartphone App | 12 Weeks Phone CBT Plus Smartphone App | Standard Diabetes Care at PCP
Number analyzed (Participants) | 3 | 2 | 3 | 2
percent adherent | 37.7 [20.2 to 56.2] | 35.7 [15.8 to 55.7] | 88.69 [79.0 to 96.1] | 84.06 [77.9 to 90.2]

4. Secondary Outcome: Diabetes Distress Scale- Change Score
Description: Levels of diabetes distress per standardized questionnaire will be measured before intervention and after intervention. Percent change of mean score between baseline and 16 weeks is reported. Adapted from Fisher, L., Glasgow, R.E., Mullan, J.T., Skaff, M.M., Polonsky, W.H. (2008) Development of a Brief Diabetes Screening Instrument. Annals of Family Medicine; 6:246-252.
Time Frame: baseline to 16 weeks
Population: Of thirteen initially randomized, one was withdrawn prior to treatment, one is missing data, and two dropped out. Therefore we do not have change scores for these pariticipants.
Measure: Mean (Full Range); unit: percent change
Arm/Group | 6 Weeks Phone CBT Plus Smartphone App | 8 Weeks Phone CBT Plus Smartphone App | 12 Weeks Phone CBT Plus Smartphone App | Treatment as Usual
Number analyzed (Participants) | 2 | 2 | 3 | 2
percent change | -17.98 [-20.4 to -15.58] | -8.33 [-37.7 to 21.1] | -40.92 [-65.3 to -1.3] | -36.22 [-39.6 to -32.8]

5. Secondary Outcome: Body Mass Index Change
Description: Change in Body Mass Index from baseline to post intervention
Time Frame: baseline to 16 weeks
Population: Of 13 initially randomized, there were 2 dropouts and one was withdrawn from the study.
Measure: Mean (Full Range); unit: kg/m^2
Arm/Group | 6 Weeks Phone CBT Plus Smartphone App | 8 Weeks Phone CBT Plus Smartphone App | 12 Weeks Phone CBT Plus Smartphone App | Treatment as Usual
Number analyzed (Participants) | 3 | 2 | 3 | 2
kg/m^2 | .23 [.1 to .3] | -1.2 [-1.3 to -1.1] | .53 [-2.2 to 2.1] | .35 [.1 to .6]

ADVERSE EVENTS:
Arm/Group | 6 Weeks Phone CBT Plus Smartphone App | 8 Weeks Phone CBT Plus Smartphone App | 12 Weeks Phone CBT Plus Smartphone App | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/4 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6 Weeks Phone CBT Plus Smartphone App (N=3) | 8 Weeks Phone CBT Plus Smartphone App (N=3) | 12 Weeks Phone CBT Plus Smartphone App (N=4) | Treatment as Usual (N=3)
concussion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — participant fell on ice when going to car and had concussion. He was removed from study due to persistent headache.

LIMITATIONS AND CAVEATS:
Pilot study with limited sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No